CLINICAL TRIAL: NCT03836573
Title: Patient Decision Aid About E-cigarettes: A Feasibility Test
Brief Title: Feasibility of a Decision Aid for E-Cigarettes in Primary Care
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Florida (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: IRB201803056; ID00023035 (Other: University of Florida); OCR19859 (Other: UF OnCore)
Record Dates: First submitted 2019-02-08; First posted 2019-02-11 (Actual); Last update posted 2019-08-22 (Actual); Status verified 2019-08

CONDITIONS: Smoking, Cigarette; Smoking Cessation
Keywords: E-cigarettes; Nicotine Replacement Therapy
MeSH Terms: conditions — Cigarette Smoking; Smoking Cessation; Vaping

STUDY DESIGN:
Intervention Model Description: The patient will answer a series of questions and based on their responses be shown information based on the group of which they are a member.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- E-cigarette only decision aid (Experimental): Patients will be provided with the Smoking Cessation iPad Decision Aid Tool consisting of information on e-cigarettes only. Patients will only be enrolled in this group in phase II if they self-identify as 'uninterested in quitting cigarettes'. During the physician encounter will be given harm-reduction guidance.
  Interventions: Behavioral: Smoking Cessation iPad Decision Aid Tool
- E-cigarette and Standard Smoking Cessation Group (Experimental): Patients will be provided with the Smoking Cessation iPad Decision Aid Tool consisting of standard smoking cessation and e-cigarette options. Patients will only be enrolled in this group in phase II if they self identify as 'interested in quitting and using e-cigarettes'. During the physician encounter will be given e-cigarette cessation guidance.
  Interventions: Behavioral: Smoking Cessation iPad Decision Aid Tool
- Standard Smoking Cessation Group (Experimental): Patients will be provided with the Smoking Cessation iPad Decision Aid Tool consisting of standard smoking cessation and e-cigarette options. All patients in phase I will be enrolled in this group. In addition, patients in phase II who self-identify as 'interested in quitting but do not use e-cigarettes' will also be enrolled in this group. During the physician encounter will be given standard smoking cessation guidance.
  Interventions: Behavioral: Smoking Cessation iPad Decision Aid Tool

INTERVENTIONS:
Behavioral: Smoking Cessation iPad Decision Aid Tool — Patients will be provided with the iPad-delivered decision aid. The patient will answer a series of questions and based on their responses be shown information based on the group of which they are a member: 1. Uninterested in quitting cigarettes (Harm-reduction Group); 2. Interested in quitting and using e-cigarettes (E-cigarette Cessation Group); 3. Interested in quitting but does not use e-cigarettes (Standard Smoking Cessation Group). Upon visiting the patient, the physician will address smoking cessation with the patient incorporating the provided decision aid results.

SUMMARY:
The study team will use a pre-post study design, in which data will be collected from 60 patients under "control" conditions (Phase I), whereby an iPad-delivered decision aid is implemented in the clinic to address only standard smoking cessation options (i.e., nicotine replacement therapy and approved prescription medications) with patients who are current smokers. After that, the iPad-delivered decision aid will be implemented with an additional 60 patients for the "intervention" condition (Phase II), whereby the decision aid will also address e-cigarettes, in addition to standard smoking cessation options.

DETAILED DESCRIPTION:
This portion of the project will take place at the UF Health Family Medicine Main Street clinic. The investigators will use a pre-post study design, in which data will be collected from 60 patients under "control" conditions (Phase I), whereby an iPad-delivered decision aid is implemented in the clinic to address only standard smoking cessation options (i.e., nicotine replacement therapy and approved prescription medications) with patients who are current smokers. After that, the iPad-delivered decision aid will be implemented with an additional 60 patients for the "intervention" condition (Phase II), whereby the decision aid will also address e-cigarettes, in addition to standard smoking cessation options. In each phase, patients visiting the clinic will be asked upon check-in to the facility if they smoke cigarettes and, if so, whether they would like to participate in research regarding smoking. Those who are interested would be directed to a research assistant in the waiting room who would present them with the study description and informed consent document, responding to any questions that they might have. Those who consent in the initial phase of the control conditions will undergo standard counseling practices their physician provides after viewing the iPad-delivered decision aid. Once the clinical visit ends, the research assistant will administer a brief survey and provide information about the two follow-up surveys, which will take place one week and 3 months after the clinical encounter.

In the intervention phase of the study (Phase II), after consenting to participate, patients will be provided with the iPad-delivered decision aid. The patient will answer a series of questions and based on their responses be shown information based on the group of which they are a member: 1. Uninterested in quitting cigarettes (harm-reduction group); 2. Interested in quitting and using e-cigarettes (e-cigarette cessation group); 3. Interested in quitting but does not use e-cigarettes (standard smoking cessation).

In both phases, after viewing the decision aid slides, patients will answer another series of questions on: value clarification; quitting readiness, interest in using e-cigarettes; interest in using other cessation methods.

Patient responses will be printed by the research assistant and provided to the nurse who is rooming the patient. While the rooming process takes place, the nurse would then place the printed decision aid paperwork in the folder outside the patient's exam room with a visual and/or verbal reminder to the physician. Upon visiting the patient, the physician would address smoking cessation with the patient incorporating the provided decision aid results. After the clinical encounter and completing check-out, the patient would return to the research assistant and conclude the experience with a short satisfaction survey that would gather information about the encounter. Participants will be followed up by preferred method (e.g., telephone, email) one week and three months after the encounter to determine changes in tobacco use perceptions and behaviors.

ELIGIBILITY:
Inclusion Criteria:

* adult smokers
* people who have smoked regular cigarettes at least once in the last month

Exclusion Criteria:

* non smokers
* pregnant women

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2019-03-06 (Actual); Primary Completion 2019-07-31 (Actual); Study Completion 2019-08-01 (Actual)

PRIMARY OUTCOMES:
Participant satisfaction with decision aid | Day 1 post visit
  A satisfaction survey will be administered to participants after the clinical encounter. Questions assess satisfaction and perceived effectiveness of the intervention.

SECONDARY OUTCOMES:
Change in cigarettes smoked per day | Baseline, Week 1, Month 3
  Change in number of cigarettes smoked per day between the groups.

CONTACTS AND LOCATIONS:
Overall Officials: Ramzi Salloum, PhD, Principal Investigator — University of Florida
Locations (1):
- UF Health at the University of Florida, Gainesville, Florida, United States

IPD SHARING:
Plan to Share IPD: No